CLINICAL TRIAL: NCT02892682
Title: The Role of the Coagulation Pathways in Recurrent Angioedema
Acronym: Angiocoag
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more inclusion
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UF 9650
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Chronic Spotaneous Urticaria, Idiopathic Non Histaminergic Angioderma, Hereditary Angioedema With C1 Inhibitor Deficiency
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 AE-Bk (Other): Arm of the recurring angiodeme medié by the bradykinine: blood test
  Interventions: Other: BLOOD TEST
- Arm 2 AE-Mast (Other): Superficial nettle rash group recurring angiodemes associated with superficial nettle rash: blood test
  Interventions: Other: BLOOD TEST
- ARM 3 AEI (Other): Arm recurring angiodemes isolate idiopathique not hostaminergique: blood test
  Interventions: Other: BLOOD TEST
- ARM 4 US (Other): Arm of superficial nettle rashes: blood test
  Interventions: Other: BLOOD TEST

INTERVENTIONS:
Other: BLOOD TEST

SUMMARY:
Previous studies reported infraclinical modifications of the homeostasis in chronic urticaria, recurrent idiopathic angioedema and hereditary angioedema. This study aim to compare groups with isolated wheals, isolated angioedema, combination of both and hereditary angioedema in terms of coagulation pathways.

DETAILED DESCRIPTION:
Previous studies reported infraclinical modifications of the homeostasis in chronic urticaria, recurrent idiopathic angioedema and hereditary angioedema. This study aim to compare groups with isolated wheals, isolated angioedema, combination of both and hereditary angioedema in terms of coagulation pathways. the main objective is to highlight a difference between the rates of different coagulation factors in the 3 groups presenting different categories of angiodemes patients with a group of patients with isolated superficial chronic urticaria

ELIGIBILITY:
Inclusion Criteria:

* recurrent angioderma

Exclusion Criteria:

* anticoagulant therapy, diseases of hemostasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Levels of several coagulation pathway markers in each group | 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No